CLINICAL TRIAL: NCT07218952
Title: Ultra-low Dose, DaT-SPECT-guided Radiation Therapy for the Treatment of Parkinson's Disease
Brief Title: Radiation Therapy (RT) for Parkinson's Disease (PD)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yasamin Sharifzadeh-Moghaddam, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-006978
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease
Keywords: anti-inflammatory; neurodegenerative disease; radiation; low-dose
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Radiation Therapy (Experimental): Patients with early-stage, non-genetic, unilateral Parkinson's Disease who will receive an ultra-low, anti-inflammatory dose of radiation therapy.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Dynamic conformal arc (DCA) therapy will be used to deliver a total of five (5) 60cGy once-a-day radiation treatments (RT) using DaT-SPECT (Dopamine Transporter-Single-Photon Emission Computed Tomography) and MRI imaging to guide radiation treatment planning.
  Other Names: LINAC TrueBeam Radiation Therapy System

SUMMARY:
The purpose of this study is to investigate the use of ultra-low, anti-inflammatory doses of radiation therapy (RT) for the treatment of Parkinson's Disease (PD). In this study, the TrueBeam LINAC utilizes a linear accelerator (LINAC) for the delivery of radiation therapy. Dynamic conformal arc (DCA) therapy will be used to deliver a total of five (5) once-a-day radiation treatments (RT) using DaT-SPECT (Dopamine Transporter-Single-Photon Emission Computed Tomography) and MRI imaging to guide radiation treatment planning.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 45 and ≤ 70 years
* Diagnosis of Parkinson's disease by a Movement Disorder Neurologist
* Confirmation of unilateral Parkinson's disease by Dopamine Transporter (DaT) scan
* A score of 2 or less on the modified Hoehn and Yahr scale
* ECOG Performance Status (PS) ≤ 2 (Appendix I).
* No known genetic causes or predisposition to Parkinson's disease or related diseases.
* Ability to complete questionnaires, neurological exam, and follow-up imaging independently or with assistance
* Ability to provide written informed consent
* Willing to provide mandatory blood samples for correlative research purposes
* Willing to return to enrolling institution for follow-up

Exclusion Criteria

* Concomitant dementia diagnosis or concerns of other memory disorder
* Parkinson's Disease medication changes within the last 3 months
* Receipt of radiation therapy for Parkinson's Disease outside Mayo Clinic, Rochester

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in progression of Parkinson's Disease | Baseline, 6 months
  Slowing of progression will be defined as a 7-point decrease in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III Motor Examination (physician-assessed motor symptoms) score. The score for this scale ranges from 0 to 132, with higher numbers indicating worse disease.

SECONDARY OUTCOMES:
Change in the Movement Disorder Society - Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS Part III) score | Baseline, 3 months, 6 months
  The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III is a physician assessed motor examination that scores symptoms on a 0-4 scale, where 0 is normal and 4 is marked severity. The total Part III score is the sum of individual item scores. Higher scores indicate a greater severity of motor deficits.
Change in Parkinson's Disease Questionnaire (PDQ-39) Score | Baseline, 3 months, 6 months
  The Parkinson's Disease Questionnaire (PDQ-39) is a 39-item questionnaire that assesses the impact of Parkinson's disease on quality of life. Each item is rated on a 5-point scale: 0: never, 1: occasionally, 2: sometimes, 3: often, and 4: always. The total score ranges from 0 (no impact) to 392 (severe impact).

CONTACTS AND LOCATIONS:
Overall Officials: Yasamin Sharifzadeh-Moghaddam, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No